CLINICAL TRIAL: NCT05174702
Title: Assessment of the Ionizing Radiation Received by the Patient and the Nursing Staff During Percutaneous or Conventional Surgery of Hallux Valgus
Brief Title: Assessment of the Ionizing Radiation Received During Percutaneous or Conventional Surgery of Hallux Valgus
Acronym: RADUS
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02408-33
Record Dates: First submitted 2021-11-30; First posted 2022-01-03 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hallux Valgus; Surgery
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Percutaneous surgery: Patient will have a percutaneous hallus valgus surgery
  Interventions: Radiation: Irradiation collected at the end of the operation on the active dosimeter
- conventional surgery: Patient will have a conventional hallus valgus surgery
  Interventions: Radiation: Irradiation collected at the end of the operation on the active dosimeter

INTERVENTIONS:
Radiation: Irradiation collected at the end of the operation on the active dosimeter — Mesure of the irradiation collected at the end of the operation on the active dosimeter for the surgeon, the patient and the operating team

SUMMARY:
To assess the average whole body radiation dose received by the surgeon, the operating team and the patient during hallux valgus surgery, depending on whether the surgery is percutaneous or conventional.

DETAILED DESCRIPTION:
Prospective, open, comparative, non-randomized, non-interventional, single-center study, focusing on two surgical strategies. Patients will be managed in accordance with current practice, the choice of surgical strategy being left to the discretion of the investigators.

Patients will be informed of the study during a preoperative visit. The data concerning them will be collected on the day of the surgery. No follow-up over time is necessary.

Passive "ring" and "cornea" dosimeters will be worn by healthcare professionals during procedures for patients included in the study. Their data will be collected each month and at the end of the study, and reported secondarily to the number of operations. Several surgeons, dressers and operating assistants will participate in the operations, their data will be aggregated taking into account their function and not individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing percutaneous or conventional hallux valgus surgery;
* Patient capable of understanding the information related to the study, of reading the information leaflet and having expressed his non-opposition to participating in the study.

Exclusion Criteria:

* Pregnant or breastfeeding woman;
* Patient under guardianship or curatorship, or under a regime of deprivation of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be managed in accordance with current practice, the choice of surgical strategy for hallus valgus (percutaneous or conventional) being left to the discretion of the investigators.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Irradiation collected at the end of the operation on the surgeon's active dosimeter | during the time of the surgery
  Measure of irradiation in mSv by a dosimeter
Irradiation collected at the end of the operation on the surgeon's active dosimeter | during the time of the surgery
  Measure of irradiation in mGy.cm² by a dosimeter

SECONDARY OUTCOMES:
Irradiation collected at the end of the operation on the patient's and operating team's | during the time of the surgery
  Measure of irradiation in mSv by a dosimeter
Irradiation collected at the end of the operation on the patient's and operating team's | during the time of the surgery
  Measure of irradiation in mGy.cm² by a dosimeter
Irradiation collected on the passive "ring" and "cornea" dosimeters of each health professional | 3 months
  Measure of irradiation in mSv by a dosimeter
Irradiation collected on the passive "ring" and "cornea" dosimeters of each health professional | 3 months
  Measure of irradiation in mGy.cm² by a dosimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Blomet, Paris, France

IPD SHARING:
Plan to Share IPD: No